CLINICAL TRIAL: NCT04511195
Title: Effectiveness and Safety of a Phytopharmaceutical Produced With an Extract of Sphaeralcea Angustifolia as a Topical Treatment of Knee Osteoarthritis: A Randomized Double Blind Clinical Trial
Brief Title: Effectiveness and Safety of Sphaeralcea Angustifolia Standardized Extract as a Topical Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sphaeralcea
Record Dates: First submitted 2020-08-05; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Knee Osteoarthritis
Keywords: Inflammation, phytopharmaceutical, outpatients, arthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Inflammation; Arthritis | interventions — Diclofenac

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the two groups: the experimental group receiving a phytopharmaceutical elaborated with the standardized extract from Sphaeralcea angustifolia, and a control group receiving an identical formulation containing Diclofenac
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both treatments present an identical appearance and are packed in white collapsible tubes, which are introduced in cardboard boxes and identified through a folio number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sphaeralcea angustifolia standardized extract (Experimental): Patients with diagnosis of knee osteoarthritis will be included in the experimental group and assigned the treatment consisting of a topical administration of a gel elaborated with the pharmaceutical formulation prepared with a standardized extract from S. angustifolia, which will be administered three times a day for four weeks.
  Interventions: Dietary Supplement: Standardized extract of Sphaeralcea angustifolia
- Diclofenac 2 % (Active Comparator): Patients with diagnosis of knee osteoarthritis will be included in the control group and assigned the treatment consisting of a topical administration of a gel elaborated with 2% diclofenac, which be administered three times a day for four weeks
  Interventions: Drug: Diclofenac Sodium Gel

INTERVENTIONS:
Dietary Supplement: Standardized extract of Sphaeralcea angustifolia — Each patient will be treated topically with a gel containing the Sphaeralcea angustifolia extract three times a day for 4 weeks. Sphaeralcea angustifolia extract is standardized in its active compounds content: Sphaeralcic acid and scopoletin
  Other Names: Sphaeralcea angustifolia standardized extract
  Arms: Sphaeralcea angustifolia standardized extract
Drug: Diclofenac Sodium Gel — Each patient will be treated topically with a gel containing 2% diclofenac three times a day for 4 weeks.
  Other Names: Diclofenac
  Arms: Diclofenac 2 %

SUMMARY:
Knee Osteoarthritis is one of the most frequent rheumatic disorders in the population and, in many cases, it causes disability due to pain, stiffness and deformation. The drugs available for treatment cause adverse events that are sometimes very severe and, for this reason, the development of new drugs for topical administration with fewer adverse events is desirable.

OBJECTIVE:

To elaborate a phytopharmaceuticals for topical administration with a standardized extract of Sphaeralcea angustifolia and evaluate its efficacy and therapeutic tolerability when administered in patients diagnosed with knee osteoarthritis.

MATERIAL AND METHODS:

An extract will be obtained from the aerial parts of the plant species S. angustifolia with which a phytomedicine will be designed in a pharmaceutical presentation for topical administration. Once the phytomedicine has been designed, it will be scaled at the pilot plant level and the drug produced will be subjected to a clinical study in order to evaluate its efficacy and therapeutic tolerability in patients diagnosed with knee osteoarthritis. Through a double-blind, randomized, controlled clinical study with 2% diclofenac, patients will be treated topically for four weeks. The evolution of the disease will be evaluated weekly during the four weeks of treatment through the Visual Analogue Scale (VAS) Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) of function. The primary outcome variable will be: therapeutic efficacy (clinical parameters for the evolution of knee pain). The secondary outcome variables will be therapeutic tolerability (side effects that are triggered by the application of the drug), and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) of function. A scale used to evaluate function of the knee

DETAILED DESCRIPTION:
In order to identify possible participants, the project will be promoted in the outpatient waiting rooms for family medicine and specialties of the General Hospital of Zone # 1 of the Mexican Institute of Social Security (IMSS) in Cuernavaca, Morelos.

People interested in participating will be asked to go to the clinical research office so that the supporting physician will perform a medical history in addition to a physical examination, in this way the clinical diagnosis of knee osteoarthritis will be made and it will be defined if the patient meets the clinical criteria necessary to be included in the study. Once it is determined that the patient is a possible candidate and the diagnostic, treatment and follow-up procedures can be continued, the patient will need to sign an informed consent letter, duly completed and authorized by the Ethics Committee. Otherwise, if patient decide not to participate, an interconsultation with the corresponding family doctor will be given.

To make the radiological diagnosis, the patient will be submitted to X-ray office, in order to take a front to back and lateral knee (s) radiograph. Once the diagnosis is corroborated, the participants will prepare a file that will contain a questionnaire with questions related to sociodemographic, personal, family and condition history, in addition, treatment will be assigned with the corresponding folio number upon admission. Each of the patients will be given oral and written instructions on how the treatment should be administered and the hygienic measures that must be followed during their participation in the study. The first administration of the treatment will be in the research office, in order to teach the participant how to do it; later, instructions about how the medication should be administered three times a day in the affected knee (s), for four weeks will be given.

Patients will be cited every week for four weeks where their evolution will be assessed; in each of the appointments. Patients will undergo a complete evaluation of their condition, there will be a format in which each of the data that is collected will be recorded, either at the interrogation or on the physical examination.

The patients will be summoned every week in order to evaluate the evolution of the disease, and consequently the therapeutic efficacy by means of the Visual Analogue Scale of pain and the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) of function, a scale used to evaluate function of the knee. The presence of adverse effects (Therapeutic tolerability) and the adherence to the treatment (based on the days of administration) will be evaluated. A concentrate related to tolerability and adherence to treatment will be filled in each of the patients.

ELIGIBILITY:
Inclusion Criteria:

* With clinical diagnosis of knee osteoarthritis based on the criteria for the classification of knee osteoarthritis and radiological classification of Kellgren and Lawrence osteoarthritis in Grade I-III.
* 40-65 years old
* Affected knee (s) must present: a) pain intensity of at least 4 cm (on the numerical scale for pain, 0-10 cm), in the knee that presents the higher pain, in the 24 hours prior to admission, b) obtain a score of not less than 50 points, according to the modified index for the clinical state of the knee with osteoarthritis, c) agree to participate in the study and sign an informed consent letter

Exclusion Criteria:

* Patients with a history of having received oral or parenteral corticosteroids for three months prior to enrollment,
* who have received anti-inflammatory drugs for 10 days before starting the study,
* who have received pain relievers for at least 3 days before the start of treatment.
* who are in some type of treatment for osteoarthritis including intra-articular infiltration.
* Patients with a Body Mass Index ≥ 30, immunosuppressed, with no controlled diabetes mellitus or hypertension
* pregnant women
* patients with high risk for not adequately managing their treatment, such as drug addicts, alcoholics
* Patients with secondary osteoarthritis (causes other than joint degeneration), with trauma to the knees in the last two months, with residual pain after trauma or post-surgery, with pain and stiffness due to tissues in the healing phase
* patients with a known intolerance to diclofenac or plant species.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-01-16 (Estimated); Study Completion 2021-06-16 (Estimated)

PRIMARY OUTCOMES:
Therapeutic efficacy: Improvement of the clinical condition higher than 80 %. It will be measured by means of Visual Analogue Scale of pain. | Four weeks
  Therapeutic efficacy will be considered when the patient presents a reduction of pain higher than 80 % on the scales of measurement Visual Analogue Scale of pain. Visual Analogue Scale (VAS) is a scale used to identify the pain intensity experienced by a patient. It consist of a line, 10 cm in length, the left side signifying no pain, and the right side signifying the worst pain: no pain (0.0 - 0.4 cm), mild pain (0.5 -4.4 cm), moderate pain (4.5 - 7.4 cm) and severe pain (7.5 - 10.0 cm).

SECONDARY OUTCOMES:
Therapeutic Tolerability: Number of patients with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events v4.0 (CTCAE v4.0) | Four weeks
  Description : Incidence and duration of adverse events monitored throughout the study by physical examination and the completion of a questionnaire. It will be considered Therapeutic Tolerability when the participant does not present adverse effect of grade 3, according to the Common Terminology Criteria for Adverse Events v 4.0
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) of function. A scale used to evaluate function of the knee | Four weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a questionnaire for the assessment of function of the affected knee. Scale describes pain in every day's life activity of the patient. Physical Function is measured by means of 17 items: using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores are summed up, with a possible score range of 0-68 for Physical Function. Higher scores on the WOMAC indicate worse functional limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Ofelia Romero-Cerecero, MD, PhD, Principal Investigator — Southern Biomedical Research Center; Susana Navarrete, Dr., Study Chair — Coordinación de Investigación en Salud
Locations (1):
- Hospital General Regional Number 1 de l IMSS en Cuernavaca, Mor., Cuernavaca, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD

REFERENCES:
- [Background] Perez-Hernandez J, Nicasio-Torres MDP, Sarmiento-Lopez LG, Rodriguez-Monroy M. Production of anti-inflammatory compounds in Sphaeralcea angustifolia cell suspension cultivated in stirred tank bioreactor. Eng Life Sci. 2019 Jan 2;19(3):196-205. doi: 10.1002/elsc.201800134. eCollection 2019 Mar. PMID 32625002
- [Background] Perez-Hernandez J, Gonzalez-Cortazar M, Marquina S, Herrera-Ruiz M, Meckes-Fischer M, Tortoriello J, Cruz-Sosa F, Nicasio-Torres Mdel P. Sphaeralcic acid and tomentin, anti-inflammatory compounds produced in cell suspension cultures of Sphaeralcea angustifolia. Planta Med. 2014 Feb;80(2-3):209-14. doi: 10.1055/s-0033-1360302. Epub 2014 Jan 31. PMID 24488717
- [Background] Romero-Cerecero O, Meckes-Fischer M, Zamilpa A, Enrique Jimenez-Ferrer J, Nicasio-Torres P, Perez-Garcia D, Tortoriello J. Clinical trial for evaluating the effectiveness and tolerability of topical Sphaeralcea angustifolia treatment in hand osteoarthritis. J Ethnopharmacol. 2013 May 20;147(2):467-73. doi: 10.1016/j.jep.2013.03.040. Epub 2013 Mar 23. PMID 23528365
- [Background] Serrano-Roman J, Nicasio-Torres P, Hernandez-Perez E, Jimenez-Ferrer E. Elimination pharmacokinetics of sphaeralcic acid, tomentin and scopoletin mixture from a standardized fraction of Sphaeralcea angustifolia (Cav.) G. Don orally administered. J Pharm Biomed Anal. 2020 May 10;183:113143. doi: 10.1016/j.jpba.2020.113143. Epub 2020 Feb 3. PMID 32045824
- [Background] Meckes M, David-Rivera AD, Nava-Aguilar V, Jimenez A. Activity of some Mexican medicinal plant extracts on carrageenan-induced rat paw edema. Phytomedicine. 2004 Jul;11(5):446-51. doi: 10.1016/j.phymed.2003.06.002. PMID 15330501